CLINICAL TRIAL: NCT05532150
Title: Conservative Versus Operative Management of First Time Shoulder Dislocations
Brief Title: Conservative Versus Operative - First Time Shoulder Dislocations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAU0965
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Shoulder Dislocation
MeSH Terms: conditions — Shoulder Dislocation | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the physical therapy (conservative) group or the operative (surgery) group if they agree to participate in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operative group (Experimental): The operative group will undergo an arthroscopic Bankart repair, which is type of surgery used to repair a dislocated shoulder.
  Interventions: Procedure: Arthroscopic Bankart repair
- Non-operative group (Active Comparator): The non-operative group will undergo physical therapy following a specific rehabilitation schedule.
  Interventions: Procedure: Physical therapy

INTERVENTIONS:
Procedure: Arthroscopic Bankart repair — Participants in this group will undergo minimally invasive surgery to repair their shoulder with a technique called a Bankart repair.
  Arms: Operative group
Procedure: Physical therapy — Participants in this group will follow a specific physical therapy rehabilitation protocol
  Arms: Non-operative group

SUMMARY:
There is no consensus regarding whether rehabilitation or surgical stabilization leads to optimized outcomes for treatment of primary anterior shoulder dislocations. This prospective, randomized controlled trial therefore aims to compare arthroscopic Bankart repair versus physical therapy for the treatment of primary anterior shoulder dislocations.

DETAILED DESCRIPTION:
While primary anterior shoulder dislocations had been previously treated conservatively, growing concerns amidst recurrent shoulder instability have fueled interest in managing these injuries with surgery to mitigate the risk of future instability events. While the significant literature investigating the rates of shoulder instability with initial operative management suggests improvement outcomes, there is limited level 1 evidence to support these implications. A randomized-controlled trial (RCT) of 21 primary anterior shoulder dislocations undergoing arthroscopic Bankart repair or rehabilitation ( 9 operative vs 12 nonoperative; mean age: 22), found lower rates of recurrent shoulder instability (11% in operative vs 72% in non-operative; p=0.004) and higher Single Assessment Numeric Evaluation (SANE) scores (88 in operative vs 57 in non-operative; p<0.002) after 36 months of follow-up. Similarly, another RCT of 76 patients (37 operative vs 39 non-operative; mean age: 22), found lower rates of recurrent shoulder instability (2.7% in operative vs 53.8% in non-operative; p<0.01) and higher Oxford assessment scores (70% with either 'excellent' or 'good' scores in operative group vs 26% with either 'excellent' or 'good' scores in non-operative group) after 10 years of follow-up. A RCT of 31 patients (16 operative vs 15 non-operative; mean age: 22), found lower rates of recurrent instability ( 19% in operative vs 60% in non-operative; p=0.02) but no significantly different Western Ontario Score Indices (WOSI) (86% in operative vs 75% in non-operative; p=0.17) at a follow up of 79 months. A RCT of 91 patients (44 operative vs 47 non-operative; mean age: 22), found lower rates of recurrent instability (2.3% in operative vs 19.1% in non-operative; p=0.01) and no significantly difference in WOSI (92.7% in operative vs 91.5% in non-operative; p>0.05) at 2 years follow-up. A RCT of 40 patients (20 operative vs 20 non-operative; mean age: 21), found lower rates of recurrent shoulder instability (10% in operative vs 70% in non-operative; p=0.0001) and a higher WOSI (17.1 in operative vs 11.5 in non-operative; p=0.035) at 2 years follow-up. The previous 5 RCT's represent the only level 1 evidence amidst a much larger proportion of lower-level evidence upon which much of the discussion of surgical vs non-operative management has been formulated. Additionally, only 2 RCT's conducted power analyses to determine if their sample size was adequate, and they did not demonstrate unanimous results with patient reported outcomes as described above. It is therefore critical to increase the amount of level 1 evidence on the topic of operative vs non-operative management of primary shoulder dislocations to better inform this debate. This study aims to compare the incidence of recurrent shoulder instability and patient reported outcomes of patients with primary anterior shoulder dislocations managed with surgery (arthroscopic Bankart repair) compared to non-operative management (standardized rehabilitation protocol, control group).

ELIGIBILITY:
Inclusion Criteria:

* patients 12 and older
* seen by the Columbia University Shoulder Elbow and Sports Medicine Service
* first time anterior shoulder dislocation diagnosis

Exclusion Criteria:

* humeral avulsion during arthroscopy
* bony defect > 25% of glenoid surface
* general anesthesia contraindication
* previous shoulder surgery
* inability or unwillingness to adhere to study participate
* lost to follow up

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2032-09 (Estimated); Study Completion 2032-09 (Estimated)

PRIMARY OUTCOMES:
Change in Western-Ontario Shoulder instability Index Score at 2 weeks | Baseline and 2 weeks
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Patient Reported Outcome Measure Information System (PROMIS) Physical function (PF) Computer Adaptive Test (CAT) at 2 weeks | Baseline and 2 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Pain Interference (PI) CAT at 2 weeks | Baseline and 2 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 2 weeks | Baseline and 2 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Western-Ontario Shoulder instability Index Score at 6 weeks | Baseline and 6 weeks
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 6 weeks | Baseline and 6 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at at 6 weeks | Baseline and 6 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 6 weeks | Baseline and 6 weeks
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Western-Ontario Shoulder instability Index Score at 3 months | Baseline and 3 months
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 3 months | Baseline and 3 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 3 months | Baseline and 3 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 3 months | Baseline and 3 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Western-Ontario Shoulder instability Index Score at 6 months | Baseline and 6 months
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 6 months | Baseline and 6 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 6 months | Baseline and 6 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 6 months | Baseline and 6 months
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Western-Ontario Shoulder instability Index Score at 1 year | Baseline and 1 year
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 1 year | Baseline and 1 year
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 1 year | Baseline and 1 year
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 1 year | Baseline and 1 year
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Western-Ontario Shoulder instability Index Score at 2 years | Baseline and 2 years
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 2 years | Baseline and 2 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 2 years | Baseline and 2 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 2 years | Baseline and 2 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Western-Ontario Shoulder instability Index Score at 5 years | Baseline and 5 years
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 5 years | Baseline and 5 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 5 years | Baseline and 5 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 5 years | Baseline and 5 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in Western-Ontario Shoulder instability Index Score at 10 years | Baseline and 10 years
  A questionnaire ranging from 0 to 2100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PF CAT at 10 years | Baseline and 10 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's physical functional capacity has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS PI CAT at 10 years | Baseline and 10 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's pain has been impacted by their shoulder injury. A lower score indicates a better outcome.
Change in PROMIS Depression CAT at 10 years | Baseline and 10 years
  A computerized questionnaire ranging from 0 to 100 points that addresses how a participant's quality of life has been impacted by their shoulder injury. A lower score indicates a better outcome.
Percentage of Participants with Recurrent Instability | 2 weeks, 6 weeks, 3 months, 6 months, 1 year, 2 years, 5 years and 10 years
  Percentage of participants in each group that experience shoulder dislocation after treatment initiates will be measured at each timepoint.

SECONDARY OUTCOMES:
Change in Constant-Murley Score at 2 weeks | Baseline and 2 weeks
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Constant-Murley Score at 6 weeks | Baseline and 6 weeks
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Constant-Murley Score at 3 months | Baseline and 3 months
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Constant-Murley Score at 6 months | Baseline and 6 months
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Constant-Murley Score at 1 year | Baseline and 1 year
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Constant-Murley Score at 2 years | Baseline and 2 years
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Constant-Murley Score at 5 years | Baseline and 5 years
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Constant-Murley Score at 10 years | Baseline and 10 years
  The Constant-Murley Score is a questionnaire that ranges from 0 (worst shoulder function) to 100 (best shoulder function) points that asks questions related to functional status and pain in the context of shoulder injuries.
Change in Subjective Shoulder Value Score at 2 weeks | Baseline and 2 weeks
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Subjective Shoulder Value Score at 6 weeks | Baseline and 6 weeks
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Subjective Shoulder Value Score at 3 months | Baseline and 3 months
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Subjective Shoulder Value Score at 6 months | Baseline and 6 months
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Subjective Shoulder Value Score at 1 year | Baseline and 1 year
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Subjective Shoulder Value Score at 2 years | Baseline and 2 years
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Subjective Shoulder Value Score at 5 years | Baseline and 5 years
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Subjective Shoulder Value Score at 10 years | Baseline and 10 years
  Single item question where participant's grade their shoulder as a percentage of their pre-injury baseline
Change in Rowe Score at 2 weeks | Baseline and 2 weeks
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Change in Rowe Score at 6 weeks | Baseline and 6 weeks
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Change in Rowe Score at 3 months | Baseline and 3 months
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Change in Rowe Score at 6 months | Baseline and 6 months
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Change in Rowe Score at 1 year | Baseline and 1 year
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Change in Rowe Score at 2 years | Baseline and 2 years
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Change in Rowe Score at 5 years | Baseline and 5 years
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Change in Rowe Score at 10 years | Baseline and 10 years
  Questionnaire that ranges from 0 (worst) of 100 (best) points that assesses stability, mobility, and function
Time to baseline functional status | Measured once per patient, depending on the time required to return to full activity (up to 10 years
  Time required to return to full activity level or return to sports after the initial injury, expressed in weeks

CONTACTS AND LOCATIONS:
Overall Officials: David P Trofa, MD, Principal Investigator — Associate Professor of Orthopaedic Surgery
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hurley ET, Manjunath AK, Bloom DA, Pauzenberger L, Mullett H, Alaia MJ, Strauss EJ. Arthroscopic Bankart Repair Versus Conservative Management for First-Time Traumatic Anterior Shoulder Instability: A Systematic Review and Meta-analysis. Arthroscopy. 2020 Sep;36(9):2526-2532. doi: 10.1016/j.arthro.2020.04.046. Epub 2020 May 8. PMID 32389771
- [Background] Bottoni CR, Wilckens JH, DeBerardino TM, D'Alleyrand JC, Rooney RC, Harpstrite JK, Arciero RA. A prospective, randomized evaluation of arthroscopic stabilization versus nonoperative treatment in patients with acute, traumatic, first-time shoulder dislocations. Am J Sports Med. 2002 Jul-Aug;30(4):576-80. doi: 10.1177/03635465020300041801. PMID 12130413
- [Background] Pouges C, Hardy A, Vervoort T, Amouyel T, Duriez P, Lalanne C, Szymanski C, Deken V, Chantelot C, Upex P, Maynou C. Arthroscopic Bankart Repair Versus Immobilization for First Episode of Anterior Shoulder Dislocation Before the Age of 25: A Randomized Controlled Trial. Am J Sports Med. 2021 Apr;49(5):1166-1174. doi: 10.1177/0363546521996381. Epub 2021 Mar 11. PMID 33705240
- [Background] Minkus M, Konigshausen M, Pauly S, Maier D, Mauch F, Stein T, Greiner S, Moursy M, Scheibel M. Immobilization in External Rotation and Abduction Versus Arthroscopic Stabilization After First-Time Anterior Shoulder Dislocation: A Multicenter Randomized Controlled Trial. Am J Sports Med. 2021 Mar;49(4):857-865. doi: 10.1177/0363546520987823. Epub 2021 Feb 17. PMID 33596092
- [Background] Jakobsen BW, Johannsen HV, Suder P, Sojbjerg JO. Primary repair versus conservative treatment of first-time traumatic anterior dislocation of the shoulder: a randomized study with 10-year follow-up. Arthroscopy. 2007 Feb;23(2):118-23. doi: 10.1016/j.arthro.2006.11.004. PMID 17276217
- [Background] Belk JW, Wharton BR, Houck DA, Bravman JT, Kraeutler MJ, Mayer B, Noonan TJ, Seidl AJ, Frank RM, McCarty EC. Shoulder Stabilization Versus Immobilization for First-Time Anterior Shoulder Dislocation: A Systematic Review and Meta-analysis of Level 1 Randomized Controlled Trials. Am J Sports Med. 2023 May;51(6):1634-1643. doi: 10.1177/03635465211065403. Epub 2022 Feb 11. PMID 35148222
- [Background] Kirkley A, Werstine R, Ratjek A, Griffin S. Prospective randomized clinical trial comparing the effectiveness of immediate arthroscopic stabilization versus immobilization and rehabilitation in first traumatic anterior dislocations of the shoulder: long-term evaluation. Arthroscopy. 2005 Jan;21(1):55-63. doi: 10.1016/j.arthro.2004.09.018. PMID 15650667